CLINICAL TRIAL: NCT03868735
Title: Evaluation of the CleanSweep™ Closed Suction System on Length of Mechanical Ventilation and Ventilator-Associated Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18110802
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CleanSweep Closed Suction System (Experimental): Device that includes balloon sweeping technology
  Interventions: Device: CleanSweep Closed Suction System
- Standard in-line suction device (No Intervention): In-line suction device already in on intubated patients with an endotracheal tube

INTERVENTIONS:
Device: CleanSweep Closed Suction System — Device with balloon sweeping technology
  Arms: CleanSweep Closed Suction System

SUMMARY:
The primary aim of this study is to evaluate the CleanSweep™ Closed Suction System on time to first successful spontaneous breathing trial in mechanically ventilated patients in the medical intensive care unit. Secondary aims of this study are to evaluate the use endotracheal tube sweeping compared to closed suctioning effect on length of mechanical ventilation, length of ICU stay, length of total hospital stay, and occurrence of ventilator-associated events.

DETAILED DESCRIPTION:
This is designed as a prospective, randomized control trial, in a large, urban, academic medical center. This study will include mechanically ventilated patients (n = 272) in the medical intensive care unit (MICU) at Rush University Medical Center. It will exclude patients with a tracheostomy on admission, those requiring extracorporeal membrane oxygenation (ECMO), or transferred from an outside facility receiving more than 24 hours of mechanical ventilation. Two groups will be randomly assigned via computer randomization. The experimental group will be placed on the CleanSweep™ Closed Suction System immediately after intubation or upon arrival to the MICU. Endotracheal tubes (ETTs) will be cleaned with the balloon sweeping technology every time a respiratory therapist suctions the patient. The control group will be placed on the standard in-line suction device. Airway suctioning will be performed in both groups as per department policy (Catheter advanced until resistance is met and withdrawn slowly for a duration no longer than 15 seconds while applying negative pressure). Both groups will also receive a ventilator bundle that consists of head of bed elevation, ETT cuff pressure management, deep vein thrombosis prevention, daily sedation interruption and SBT, and oral care every 4 hours with chlorhexidine at 12pm (noon) and 12am midnight.

ELIGIBILITY:
Inclusion Criteria:

* Orally intubated patient with endotracheal tube
* Mechanically ventilated less than 24 hours prior to enrollment

Exclusion Criteria:

* Less than 18 years old
* Tracheostomy tube
* Extracorporeal membrane oxygenation
* Transfer from outside hospital with more than 24 hours of mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B Scott, MSc, Principal Investigator — Rush University University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Started | 136 | 136
Completed | 136 | 136
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 63 [52 to 72] | 63 [52 to 74] | 63 [52 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 71 | 129
  Male | 78 | 65 | 143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 57 | 51 | 108
  Caucasian | 36 | 30 | 66
  Hispanic | 31 | 44 | 75
  Asian | 4 | 5 | 9
  Other | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 136 | 136 | 272
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.8 [24 to 34] | 29.3 [25 to 35] | 29.05 [24.5 to 34.5]

OUTCOME MEASURES:

1. Primary Outcome: Length of Time on a Mechanical Ventilator
Description: Length of time on mechanical ventilation was recorded in hours.
Time Frame: Hospital admission to discharge (up to about 20 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Number analyzed (Participants) | 136 | 136
hours | 70.6 [37 to 148] | 72.2 [37 to 187]

2. Secondary Outcome: Time to First Successful Spontaneous Breathing Trial (SBT)
Description: Time to first successful SBT in mechanically ventilated patients in the medical intensive care unit.
Time Frame: Hospital admission to discharge (up to about 20 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Number analyzed (Participants) | 136 | 136
hours | 45.7 [27 to 95] | 46.7 [30 to 87]

3. Secondary Outcome: Length of Time in the Intensive Care Unit
Description: Length of time spent in the intensive care units in days
Time Frame: Hospital admission to discharge (up to about 20 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Number analyzed (Participants) | 136 | 136
days | 7.8 [4 to 18] | 9 [4 to 20]

4. Secondary Outcome: Length of Total Hospital Stay
Description: Length of total time spent in the hospital in days
Time Frame: Hospital admission to discharge (up to about 20 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Number analyzed (Participants) | 136 | 136
days | 13.9 [8 to 25] | 14.7 [8 to 26]

5. Secondary Outcome: Number of Participants With Ventilator-associated Events
Description: Number of Participants with ventilator-associated events, like pneumonia
Time Frame: Hospital admission to discharge (up to about 20 days)
Measure: Number; unit: participants
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
Number analyzed (Participants) | 136 | 136
participants | 16 | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CleanSweep Closed Suction System | Standard In-line Suction Device
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/136
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/136
Other Adverse Events (participants affected / at risk) | 0/136 | 0/136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT03868735/Prot_SAP_001.pdf